CLINICAL TRIAL: NCT01372293
Title: 17-hydroxysteroid Dehydrogenase Type 5 Gene Polymorphism (71A/G HSD17B5 SNP) and Effects of Oral Contraceptive Pill on Hirsutism, Androgens and Metabolic Profile in Non-obese PCOS Women: a Pilot Study
Brief Title: 71A/G HSD17B5 SNP and Effects of Oral Contraceptive Pill in PCOS Women
Acronym: 17b-ACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Denusa Wiltgen, MD,PhD, Federal University of Rio Grande do Sul
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-245
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; oral contraceptive pill; polymorphisms
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oral contraceptive pill — ethinyl oestradiol 20ug plus gestodene 75ug during 6 cycles

SUMMARY:
An association of the single nucleotide polymorphism (SNP) in the promoter gene that codify for 17b-HSD5 enzyme (71A>G) with polycystic ovary syndrome (PCOS) and hyperandrogenemia has been suggested in previous studies.

Given the role of 17b-HSD5 in androgenic metabolism producing testosterone from precursors, the investigators hypothesis is that women with PCOS and with the variant allele G have a poor response on hirsutism and on hormonal and metabolic variables after oral contraceptive pill (OCP) treatment for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* hirsute women with polycystic ovary syndrome

Exclusion Criteria:

* Use of any drugs known to interfere with hormone levels for at least 3 months before the study
* Women with type 2 diabetes, homa index > 3.8, liver or renal disease or thyroid dysfunction
* Other hyperandrogenic disorders than PCOS

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes at Ferriman- Gallwey score | 6 months

SECONDARY OUTCOMES:
Changes at testosterone levels | 6 months
Changes in lipid profile | 6 months

REFERENCES:
- [Derived] Maier PS, Mattiello SS, Lages L, Spritzer PM. 17-Hydroxysteroid dehydrogenase type 5 gene polymorphism (-71A/G HSD17B5 SNP) and treatment with oral contraceptive pills in PCOS women without metabolic comorbidities. Gynecol Endocrinol. 2012 Aug;28(8):606-10. doi: 10.3109/09513590.2011.650760. Epub 2012 Feb 14. PMID 22329763